CLINICAL TRIAL: NCT07161427
Title: Biomechanics-based Fu's Subcutaneous Needling Versus Bracing Combined With Resistance Training in the Treatment of Postacute Lateral Ankle Sprain and the Prevention of Chronic Ankle Instability: A Randomized Controlled Trial Protocol
Brief Title: Fu's Subcutaneous Needling for Postacute Lateral Ankle Sprain and Prevention of Chronic Ankle Instability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Lingjing Chen, Principal Investigator, Guangzhou University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YF 2025 -158-01
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Chronic Ankle Instability; Lateral Ankle Sprain
Keywords: Fu's subcutaneous needling; Ankle sprain; Postacute lateral ankle sprain; Chronic ankle instability; Functional rehabilitation; Balance; Non-surgical therapy
MeSH Terms: conditions — Ankle Injuries | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: To maximally reduce other potential sources of bias, the intervention operators, outcome assessors, data collectors, and data analysts act as independent researchers. Except for the intervention operators, the researchers should not be aware of the participants' group assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FSN group (Experimental): Participants first assume the supine position. After routine disinfection, the Fu's subcutaneous needle is inserted parallelly into the subcutaneous loose connective tissue around the pathologically taut muscles (such as the tibialis anterior, peroneus longus, gastrocnemius, soleus, peroneus brevis, and extensor digitorum longus, etc.). After the needle is fully inserted, fix the protruding part of the hose holder onto the card slot.To minimize the participants' perception of pain, the doctor uses the index finger and ring finger to perform a smooth, gentle, and fan-shaped swinging motion in an alternating front-to-back manner.The sector angle is approximately 60°. It makes a total of round - trips 45 times within 30 seconds. The rocking motion is accompanied by Reperfusion Approach: A set of procedures consists of 20 times of rocking followed by 10 seconds of reperfusion method. Each target lesioned tense muscle requires 2 - 3 sets of the above - mentioned procedures.
  Interventions: Procedure: Fu's Subcutaneous Needling therapy
- combined treatment group (Active Comparator): Participants in the combination therapy group wore ankle orthoses during their daily activities from 9:00 to 20:00 every day for a total of 2 weeks. During the treatment with ankle joint orthosis, complete the resistance training every day.
  Interventions: Behavioral: Ankle joint aids combined with exercise therapy

INTERVENTIONS:
Procedure: Fu's Subcutaneous Needling therapy — Participants first assume the supine position. After routine disinfection, the Fu's subcutaneous needle is inserted parallelly into the subcutaneous loose connective tissue around the pathologically taut muscles (such as the tibialis anterior, peroneus longus, gastrocnemius, soleus, peroneus brevis, and extensor digitorum longus, etc.). After the needle is fully inserted, fix the protruding part of the hose holder onto the card slot.To minimize the participants' perception of pain, the doctor uses the index finger and ring finger to perform a smooth, gentle, and fan-shaped swinging motion in an alternating front-to-back manner.The sector angle is approximately 60°. It makes a total of round - trips 45 times within 30 seconds. The rocking motion is accompanied by Reperfusion Approach: A set of procedures consists of 20 times of rocking followed by 10 seconds of reperfusion method. Each target lesioned tense muscle requires 2 - 3 sets of the above - mentioned procedures.
  Arms: FSN group
Behavioral: Ankle joint aids combined with exercise therapy — Participants in the combination therapy group wore ankle orthoses during their daily activities from 9:00 to 20:00 every day for a total of 2 weeks. To ensure standardization, a unified specification is selected for the ankle joint orthosis: Product number: 100159548, the 195R Super Sports Ankle Brace for Inversion/Eversion Sprains and Ligament Fixation by McDavid from the United States. During the treatment with ankle joint orthosis, complete the resistance training every day.
  Arms: combined treatment group

SUMMARY:
Introduction: Fu's Subcutaneous Needling (FSN) is a new type of acupuncture treatment method based on the subcutaneous tissue sweeping technique, and it has been proven to have a good therapeutic effect on ankle sprain. However, at present, the difference between its curative effect and the ankle joint orthosis and exercise therapy recommended by the Guidelines remains unclear. Therefore, this study aims to explore the improvement effects of FSN on pain relief, joint function improvement, and ankle balance ability by comparing with ankle orthosis combined with exercise therapy. Verify whether it is more helpful in preventing the progression of lateral ankle sprain (LAS) to chronic ankle instability (CAI) and provide evidence-based basis for clinical decision-making.

Methods and analysis: This study is a randomized, parallel - controlled, single - center prospective clinical study. This study will include 60 subjects with postacute lateral ankle sprain and divide them into the FSN group and the combined treatment group. There are 30 cases in each group. The FSN group will be treated with Fu's subcutaneous needling three times a week for a total of two weeks. The Combined treatment group will wear ankle orthotics from 9:00 to 20:00, and complete resistance exercise training every day for a total of two weeks.Patients will be followed up for 6 months after the treatment. The main efficacy index is the change value of the Visual Analog Scale (VAS) compared to the baseline after 2 weeks of treatment. The secondary indicators include active range of motion (ROM) of the ankle joint, Star Excursion Balance Test (SEBT), and the Foot and Ankle Ability Measure (FAAM) to prove the clinical efficacy.

Ethics and dissemination: This study strictly adheres to the ethical guidelines of the Declaration of Helsinki.This study has passed the review of the Ethics Committee of Guangdong Provincial Hospital of Chinese Medicine. Approval No.: YF 2025 - 158 - 01. All subjects will sign a written informed consent form. The research results will be publicly published in journals indexed by SCI.

Keywords: Fu's subcutaneous needling, Ankle sprain, Postacute lateral ankle sprain, Chronic ankle instability, Functional rehabilitation, Balance, Non-surgical therapy

ELIGIBILITY:
Inclusion Criteria:

1. Patients with first-time lateral ankle sprains
2. The patient presents with symptoms of swelling and aching and weakness in the ankle joint. There may be a feeling of friction during joint movement, and the symptoms are aggravated after long - distance walking or on rainy and overcast days.
3. The patient presents with swelling and tenderness in the anteroinferior aspect of the lateral malleolus and the anterolateral aspect of the medial malleolus, and has limited mobility during inversion and flexion-extension.
4. Auxiliary examinations: No fracture or dislocation was found in the patient during the examination, and no fracture was detected by X-ray examination.
5. The patient's sprain time is more than 3 weeks and within 6 months.
6. Those who have not received surgical treatment at other medical institutions before coming to our hospital for treatment, can complete the treatment and accept follow - up.
7. The patients' ages range from 18 to 60 years old.
8. The patient voluntarily and is capable of signing the Informed Consent Form.

Exclusion Criteria:

1. Those with complete rupture of fractures or soft tissues such as muscles, tendons, and ligaments
2. Patients with severe primary diseases such as heart, liver, kidney, hematopoietic system diseases and mental diseases
3. Patients with tumors or tuberculosis in the ankle joint
4. Patients with rheumatic and rheumatoid arthritis, or gout.
5. Patients with acute inflammatory reactions such as redness, swelling, heat and pain and signs of infection in the ankle joint, or those accompanied by severe osteoarthritis.
6. Patients with abnormal coagulation function or bleeding tendency, such as those with thrombocytopenia and severe diabetes.
7. Patients during pregnancy and lactation
8. Patients with damaged skin at the necessary needle insertion sites.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | The evaluators measure the outcomes at the baseline, on day 7, day 14, and during the follow - up period (day 28, day 42, 3 months, and 6 months after the start of treatment).
  The scoring range of the Visual Analogue Scale (VAS) is 0 - 100 mm, which is used for objectively quantifying the pain level. The participants were instructed to indicate the severity of their ankle pain by marking a point on a continuous horizontal line segment, with 0 mm representing the least pain and 100 mm representing the most severe pain.

SECONDARY OUTCOMES:
active range of motion of the ankle joint | was measured at the baseline, on the 14th day, and during the follow - up period.
  Active range of motion (ROM), including plantar flexion, dorsiflexion, inversion and eversion, was measured at the baseline, on the 14th day, and during the follow - up period.
The Star Excursion Balance Test | at the baseline, on the 7th day, on the 14th day, and during the follow-up period.
  The Star Excursion Balance Test (SEBT) has sufficient sensitivity and high test-retest reliability in the ankle dynamic balance test.
The Foot and Ankle Ability Measure | at the baseline, on the 14th day, and during the follow - up period.
  The Foot and Ankle Ability Measure (FAAM) is a self - assessment scale commonly used for the individual physical function in injuries related to the foot and ankle joint, which is completed by patients. It includes two subscales: Foot and Ankle Ability Measure - Activity of Daily Living (FAAM - ADL) and Foot and Ankle Ability Measure - Sports (FAAM - S). FAAM - ADL (84 points): It covers 21 daily activities such as standing, walking, squatting, standing on tiptoe, walking for different durations, and doing housework. FAAM - S (32 points): It includes 8 sports - related activities such as running, jumping take - off, landing after a jump, and starting or ending a run. The score range of both sub - scales is 0 - 100%. A total score ≥ 80% indicates a satisfactory functional level, and < 80% indicates functional limitation.
Cumberland Ankle Instability Tool | at the baseline, on the 14th day, and during the follow - up period.
  CAIT consists of 9 items, with scores ranging from 0 to 30. The lower the score, the worse the ankle stability. The threshold for identifying people with chronic ankle instability is inconsistent in different language versions. A score of less than 24 in the Chinese version of CAIT is diagnosed as chronic ankle instability. It is measured at baseline, 14 th and 6 th month follow-up.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Pierobon A, Raguzzi I, Solino S, Salzberg S, Vuoto T, Gilgado D, Perez Calvo E. Minimal detectable change and reliability of the star excursion balance test in patients with lateral ankle sprain. Physiother Res Int. 2020 Oct;25(4):e1850. doi: 10.1002/pri.1850. Epub 2020 May 26. PMID 32458531
- [Background] Goulart Neto AM, Maffulli N, Migliorini F, de Menezes FS, Okubo R. Validation of Foot and Ankle Ability Measure (FAAM) and the Foot and Ankle Outcome Score (FAOS) in individuals with chronic ankle instability: a cross-sectional observational study. J Orthop Surg Res. 2022 Jan 21;17(1):38. doi: 10.1186/s13018-022-02925-9. PMID 35062990
- [Background] de Noronha M, Refshauge KM, Herbert RD, Kilbreath SL, Hertel J. Do voluntary strength, proprioception, range of motion, or postural sway predict occurrence of lateral ankle sprain? Br J Sports Med. 2006 Oct;40(10):824-8; discussion 828. doi: 10.1136/bjsm.2006.029645. Epub 2006 Aug 18. PMID 16920769
- [Background] Hiller CE, Refshauge KM, Bundy AC, Herbert RD, Kilbreath SL. The Cumberland ankle instability tool: a report of validity and reliability testing. Arch Phys Med Rehabil. 2006 Sep;87(9):1235-41. doi: 10.1016/j.apmr.2006.05.022. PMID 16935061